CLINICAL TRIAL: NCT04061304
Title: A Clinical Trial Into the Efficacy of rTMS Treatment for Treating Anorexia Nervosa and Bulimia Nervosa
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Challenges with funding acquisition prevented study commencement.
Sponsor: University of Manitoba (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HS22828 (B2019:033)
Record Dates: First submitted 2019-07-02; First posted 2019-08-19 (Actual); Last update posted 2021-10-08 (Actual); Status verified 2021-03

CONDITIONS: Eating Disorders; Anorexia Nervosa; Bulimia Nervosa
Keywords: rTMS
MeSH Terms: conditions — Feeding and Eating Disorders; Anorexia Nervosa; Bulimia Nervosa | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Active rTMS (Anorexia Nervosa) (Experimental): Patients in this arm will receive 40 sessions of active rTMS. Every day, the first session of rTMS for both groups will be applied to the left DLPFC using intermittent Theta Burst Stimulation (iTBS).
  For the second session each day the patients in the anorexia group will receive low-frequency treatment (1 Hz, 60 second cycles, 30 second inter-train interval, 20 trains, 1200 total pulses) at 120% of the resting motor threshold to the orbitofrontal cortex
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation
- Active rTMS (Bulimia Nervosa) (Experimental): Patients in this arm will receive 40 sessions of active rTMS. Every day, the first session of rTMS for both groups will be applied to the left DLPFC using intermittent Theta Burst Stimulation (iTBS).
  For the second session each day the patients in the bulimia group will receive high-frequency (10 Hz, 5 second cycles, 50 pulses, 25 second inter-train interval, 60 trains, 3000 total) at 120% of the resting motor threshold treatment to the left dorsomedial prefrontal cortex
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation
- Sham rTMS (Anorexia Nervosa) (Sham Comparator): Patients in this arm will receive 40 sessions of sham rTMS. They will be set up the same as the active Anorexia Nervosa group however their will be no actual brain stimulation.
  Interventions: Device: Sham Transcranial Magnetic Stimulation
- Sham rTMS (Bulimia Nervosa) (Sham Comparator): Patients in this arm will receive 40 sessions of sham rTMS. They will be set up the same as the active Bulimia Nervosa group however their will be no actual brain stimulation.
  Interventions: Device: Sham Transcranial Magnetic Stimulation

INTERVENTIONS:
Device: Repetitive Transcranial Magnetic Stimulation — A non-invasive method of brain stimulation.
  Arms: Active rTMS (Anorexia Nervosa); Active rTMS (Bulimia Nervosa)
Device: Sham Transcranial Magnetic Stimulation — A device designed to look, sound, and feel like a real magnetic stimulation coil without actually stimulating the brain.
  Arms: Sham rTMS (Anorexia Nervosa); Sham rTMS (Bulimia Nervosa)

SUMMARY:
This is a pilot study to test the efficacy of repetitive transcranial magnetic stimulation (rTMS) in treating individuals with Anorexia Nervosa and Bulimia Nervosa. The main objective of this study is to determine the short and long-term efficacy of repetitive transcranial magnetic stimulation (rTMS) in reducing eating disorder symptoms (i.e. binging, purging, restricting, intense fear of gaining wait, etc;) in Anorexia Nervosa and Bulimia Nervosa.

The investigators will also be comparing the brain activity patterns of individuals with Anorexia Nervosa and Bulimia Nervosa to healthy controls using electroencephalography (EEG). Further, the investigators would like to examine if the activation patterns in these patients change after receiving rTMS.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of Anorexia Nervosa or Bulimia Nervosa, must pass rTMS screening questionnaire

Exclusion Criteria:

* Diagnosis of another psychiatric disorder, except MDD.
* Any rTMS counter-indications:
* History of seizures
* Metal in head
* Currently pregnant
* Having received rTMS for any reason in the past as this would interfere with participant blinding.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2021-03-19 (Actual); Study Completion 2021-03-19 (Actual)

PRIMARY OUTCOMES:
Weekly Binge/Purge Frequency on Eating Disorder Examination | baseline, after week 1, week 2, and week 3 of treatment, 3 months post treatment, and 6 months post treatment.
  Outcome measured by change of binge/purge episodes from baseline to the end of treatment. If the participant has a final score of 0 binges and 0 purges they will be considered in remission. A 50% improvement will be defined as a response to the rTMS.

SECONDARY OUTCOMES:
Change in Beck Anxiety Inventory (BAI) | baseline, after week 1, week 2, and week 3 of treatment, 3 months post treatment, and 6 months post treatment.
  Outcome range: 0-63, with higher scores reflecting higher levels of anxiety. A total of 21 questions are summed for a total score out of 63.
Change in Beck Depression Inventory (BDI) | baseline, after week 1, week 2, and week 3 of treatment, 3 months post treatment, and 6 months post treatment.
  Outcome range: 0-63, with higher scores reflecting higher levels of depression. A total of 21 questions are summed for a total score out of 63.

CONTACTS AND LOCATIONS:
Overall Officials: Mandana Modirrousta, MD PhD FRCPC, Principal Investigator — University of Manitoba